CLINICAL TRIAL: NCT04109105
Title: Prospective Pilot Study for the Efficacy and Security Analysis in the Protection of Ileocolic Anastomosis Conducted in Laparoscopic Right Hemicolectomy Because of Colon Cancer, Using a Using a NHS-PEG (N-hydroxysuccinimide Functionalized Polyethylene Glycol) Coated Collagen Patch.
Brief Title: Study for the Efficacy and Security Analysis in the Protection of Ileocolic Anastomosis Conducted in Laparoscopic Right Hemicolectomy Because of Colon Cancer, Using a NHS-PEG Coated Collagen Patch.
Acronym: ANASTOPATCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-HEMOPATCH-2018-02
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Adenocarcinoma Colon
Keywords: Colon neoplasia; Ascendant colon; Surgical anastomosis; Anastomotic leak; Collagen; Polyethylene glycol; Hemopatch
MeSH Terms: conditions — Colonic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NHS-PEG coated collagen patch cohort: Patients diagnosed of colon adenocarcinoma that have ileocolic anastomosis after undergoing a laparoscopic right hemicolectomy surgery.
  Interventions: Other: NHS-PEG coated collagen patch

INTERVENTIONS:
Other: NHS-PEG coated collagen patch — Analysis of the number and seriousness of leaks in the ileocolic anastomosis after using a NHS-PEG coated collagen patch reinforcement.
  Other Names: Hemopatch

SUMMARY:
The aim of this study is to analyse the effectiveness and security in the prevention of anastomotic leakage by protecting the ileocolic anastomosis with a reabsorbable NHS-PEG collagen patch.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Ability to understand and make their own decision to participate in the study.
* Pre-surgery right colon adenocarcinoma pathological diagnosis.
* Patient with a mechanic, intra or extracorporeal ileocolic anastomosis.

Exclusion Criteria:

* Urgent intervention.
* Simultaneous colon cancer.
* M1 pre-surgery staging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a programmed right laparoscopic hemicolectomy for right colon adenocarcinoma with curative intention at the Virgen Macarena University Hospital during the necessary period of time to achieve the proposed number of patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and security analysis in the prevention of anastomosis leakage through the protection of ileocolic anastomosis with NHS-PEG coated collagen patch. | Up to 30 days after the surgery
  Ileocolic anastomosis leakage existence of evidence and seriousness.

SECONDARY OUTCOMES:
Analysis of the percentage of leaks in the ileocolic anastomosis reinforced with NHS-PEG coated collagen patch. | Up to 30 days after the surgery
  Percentage of leaks that occur in the ileocolic anastomosis after being reinforced with NHS-PEG coated collagen patch.
Number of complications related to anastomotic leakage in patients with ileocolic anastomosis reinforced with NHS-PEG coated collagen patch. | Up to 30 days after the surgery
  Number and type of complications due to the anastomotic leakage in patients with ileocolic anastomosis reinforced with NHS-PEG coated collagen patch.
Number of surgical repetitions. | Up to 30 days after the surgery
  Number of following surgeries that the patient has to undergo due to the failure of the collagen patch ileocolic anastomosis protection.
Number of hospital readmissions. | Up to 30 days after the surgery
  Number of times that the patient has to be rehospitalized due to the failure of the collagen patch ileocolic anastomosis protection.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Gómez Rosado, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain